CLINICAL TRIAL: NCT00749008
Title: Early Prediction of Cerebral Palsy in Preterm Infants and Term Infants Using Detection of Generalized Movements
Brief Title: Study of Generalized Movements for Early Prediction of Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Charles R. Neal, (Other)
Collaborators: Hawaii Community Foundation (Other)
Responsible Party: Sponsor-Investigator, Charles R. Neal,, Principal Investigator, Hawaii Pacific Health
Organization: Hawaii Pacific Health (Other)
Other Study IDs: RP#07-130-1-HPH1
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cerebral Palsy; Prematurity
Keywords: Cerebral palsy; Generalized movements; Fidgety movements; Prechtl
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Term Infants: High risk infants with history of respiratory insufficiency requiring NICU care.
- Preterm Infants: Infants less than 37 weeks gestational age.

SUMMARY:
The purpose of this study is to assess the predictive value of generalized movements in preterm and term infants who are at risk for development of cerebral palsy. The investigators will identify at-risk infants and observe their generalized movements, conduct a two year longitudinal follow-up, and interpret the predictive value of the investigators assessments based on the diagnosis of cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is considered a clinical syndrome caused by a preceding brain injury early in brain development that results in static neurological deficits. These deficits usually involve the somatomotor system manifesting as hemi-, di- or quadriplegia. Cerebral palsy can also manifest as hypertonicity and contractures, sensory deficits, hearing and visual difficulties, feeding problems and global developmental delay and almost always coincides with chronic lung disease. The most common causes of cerebral palsy are hypoxic-ischemic brain injury, periventricular leukomalacia or intraventricular and/or parenchymal hemorrhage that occurs in the first year of life. Hypoxic brain injury as a result of poor oxygen delivery often occurs in the perinatal period but can also be caused by pulmonary dysfunction. Thus, pulmonary diseases such as bronchopulmonary dysplasia, pneumonia, meconium aspiration syndrome, congenital diaphragmatic hernia and respiratory distress syndrome can lead to hypoxic brain injury and consequent CP. Less common etiologies are genetic disorders, infections and intrapartum injuries. Current treatments of CP are targeted to maintaining function, relieving contractures, improving nutrition and providing developmental supportive care, but to date there is no cure or preventive guideline. Moreover, supportive measures and family counseling is delayed since CP can be diagnosed only at the age of 18-24 months. As a result, interventions that may aid in limiting CP effects are delayed due to the lack of a predictive diagnostic assessment during the first six months of life. Head ultrasound, EEG and functional MRI have been tested for their predictive value before the actual diagnosis of cerebral palsy. The low sensitivity of these studies shows that they are not useful as screening tools. Heinz Prechtl, an Austrian neurologist, developed a clinical assessment method to study the spontaneous movements of preterm and term infants. Monitoring of cramped synchronized generalized movements and fidgety movements has resulted in 100% sensitivity and 95% specificity in predicting cerebral palsy in many studies. A meta-analysis of predictive tools for cerebral palsy identified Prechtl's method as superior to head ultrasound or MRI. These studies have not been repeated in the USA. Our aim is to assess the predictive value of Prechtl's method in Hawaii, in preterm and term infants with and without lung disease, who are at risk for development of cerebral palsy. We will compare the incidence of pulmonary diseases and cerebral palsy and observe any relationship between the development of lung disease and brain injury. We will identify at risk infants and observe their generalized movements according to Prechtl's assessment. We will conduct a 2-year longitudinal follow up of our patients and interpret the predictive value of our assessment based on the diagnosis of cerebral palsy. We will compare the sensitivity and positive predictive value of head ultrasound and the assessment of generalized movements. It is hoped that this assessment will allow us to start supportive measures at an earlier stage of life, thus improving the outcome of children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns with pulmonary diseases (meconium aspiration, congenital diaphragmatic hernia, bronchopulmonary dysplasia, pneumonia, lobar emphysema and respiratory distress syndrome)
* Preterm infants less than 30 weeks of gestational age or less than 1500g weight
* Preterm or term infants with intrauterine growth retardation
* Infants with the diagnosis of IVH larger than grade II
* Infants diagnosed with periventricular leukomalacia
* Any preterm and term infant who experienced hypoxic-ischemic injury, defined as having a 5 minute Apgar score less than 4 or requiring resuscitation >10 minutes.

Exclusion Criteria:

* Congenital anomalies
* Congenital heart disease
* Any genetic anomalies

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm and term infants in the state of Hawaii, with and without lung disease, who are at risk for development of cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2008-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Cerebral Palsy | Two Years of Age

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Neal, MD, PhD, Principal Investigator — University of Hawaii
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States